CLINICAL TRIAL: NCT04608513
Title: A Single-center, Double-blind, Randomized, Placebo-controlled Phase 1 Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Single- and Multiple-ascending Doses of ACT-1014-6470 in Healthy Subjects
Brief Title: A Placebo-controlled Phase 1 Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Single- and Multiple-ascending Doses of ACT-1014-6470 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-087-102
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Healthy
MeSH Terms: interventions — ACT-1014-6470

STUDY DESIGN:
Intervention Model Description: Single-center, double-blind, randomized, placebo-controlled, single- and multiple-ascending dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- ACT-1014-6470 single dose (dose level 1) (Experimental): Soft capsule for oral administration
  Interventions: Drug: ACT-1014-6470
- Placebo single dose (dose level 1) (Placebo Comparator): Soft capsule for oral administration
  Interventions: Drug: Placebo
- ACT-1014-6470 single dose (dose level 2) (Experimental): Soft capsule for oral administration
  Interventions: Drug: ACT-1014-6470
- Placebo single dose (dose level 2) (Placebo Comparator): Soft capsule for oral administration
  Interventions: Drug: Placebo
- ACT-1014-6470 multiple dose (dose level 1) (Experimental): Soft capsule for oral administration
  Interventions: Drug: ACT-1014-6470
- Placebo multiple dose (dose level 1) (Placebo Comparator): Soft capsule for oral administration
  Interventions: Drug: Placebo
- ACT-1014-6470 multiple dose (dose level 2) (Experimental): Soft capsule for oral administration
  Interventions: Drug: ACT-1014-6470
- Placebo multiple dose (dose level 2) (Placebo Comparator): Soft capsule for oral administration
  Interventions: Drug: Placebo
- ACT-1014-6470 multiple dose (dose level 3) (Experimental): Soft capsule for oral administration
  Interventions: Drug: ACT-1014-6470
- Placebo multiple dose (dose level 3) (Placebo Comparator): Soft capsule for oral administration
  Interventions: Drug: Placebo
- ACT-1014-6470 multiple dose (dose level 4) (Experimental): Soft capsule for oral administration
  Interventions: Drug: ACT-1014-6470
- Placebo multiple dose (dose level 4) (Placebo Comparator): Soft capsule for oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-1014-6470 — Soft capsules for oral administration
  Arms: ACT-1014-6470 multiple dose (dose level 1); ACT-1014-6470 multiple dose (dose level 2); ACT-1014-6470 multiple dose (dose level 3); ACT-1014-6470 multiple dose (dose level 4); ACT-1014-6470 single dose (dose level 1); ACT-1014-6470 single dose (dose level 2)
Drug: Placebo — Soft capsules for oral administration
  Arms: Placebo multiple dose (dose level 1); Placebo multiple dose (dose level 2); Placebo multiple dose (dose level 3); Placebo multiple dose (dose level 4); Placebo single dose (dose level 1); Placebo single dose (dose level 2)

SUMMARY:
A safety and tolerability study in healthy subjects including examination of how the body takes up, distributes, and gets rid of ACT-1014-6470

ELIGIBILITY:
Inclusion Criteria:

General criteria

* Signed informed consent prior to any study-mandated procedure.
* Healthy male subjects (both study parts) and female subjects of nonchildbearing potential (Part B) aged between 18 and 55 years (inclusive) at Screening.
* Healthy on the basis of medical history, physical examination, cardiovascular assessments, and clinical laboratory tests.
* Male subjects with a partner that might become pregnant must either be vasectomized or agree to practice adequate contraception from admission to the study site until 3 months after dosing, or the partner must consistently and correctly use (from Screening, during the entire study, and for at least 3 months after last study treatment intake) a highly effective method of contraception.

Criteria for Part B only:

• Women of non-childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day-1.

Exclusion Criteria:

* Previous exposure to the study medication.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which, in the opinion of the investigator, are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment.
* Relevant bacterial, viral, fungal, or protozoal infection that manifested within the last 6 weeks prior to Screening and/or ongoing relevant bacterial, viral, fungal, or protozoal infection, as judged by the investigator, and/or evidence of immune dysfunction based on laboratory tests at Screening.
* Any signs or symptoms of active, ongoing infection judged to be clinically relevant by the investigator (special attention should be given to clinical signs and symptoms consistent with COVID-19, e.g., fever, dry cough, dyspnea, sore throat, or fatigue).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Safety profile including incidence of treatment-emergent adverse events. | Safety and tolerability assessments will be performed at predefined time points from Day 1 to Day 4 in Part A and Day 1 to Day 10 in Part B (total duration: max. 50 days).

SECONDARY OUTCOMES:
Part A - Single ascending dose (SAD): Area under the plasma concentration-time curve (AUC) from zero to time t of the last measured concentration above the limit of quantification (AUC0-t). | Blood samples for the determination of the PK parameters will be collected at predefined time points from Day 1 to Day 4 (total duration: max. 4 days).
Part A - Single ascending dose (SAD): Area under the plasma concentration-time curve (AUC) from zero to infinity (AUC0-inf). | Blood samples for the determination of the PK parameters will be collected at predefined time points from Day 1 to Day 4 (total duration: max. 4 days).
Part A - Single ascending dose (SAD): Maximum plasma concentration (Cmax). | Blood samples for the determination of the PK parameters will be collected at predefined time points from Day 1 to Day 4 (total duration: max. 4 days).
Part A - Single ascending dose (SAD): Time to reach Cmax (tmax). | Blood samples for the determination of the PK parameters will be collected at predefined time points from Day 1 to Day 4 (total duration: max. 4 days).
Part A - Single ascending dose (SAD): Terminal half-life (t½). | Blood samples for the determination of the PK parameters will be collected at predefined time points from Day 1 to Day 4 (total duration: max. 4 days).
Part B - Multiple ascending dose (MAD): AUC during a dosing interval (AUCτ) following the first and the last dose. | Blood samples for the determination of the PK parameters will be collected at predefined time points from Day 1 to Day 10 (total duration: max. 10 days).
Part B - Multiple ascending dose (MAD): Cmax of the first and the last dosing interval. | Blood samples for the determination of the PK parameters will be collected at predefined time points from Day 1 to Day 10 (total duration: max. 10 days).
Part B - Multiple ascending dose (MAD): tmax of the first and the last dosing interval. | Blood samples for the determination of the PK parameters will be collected at predefined time points from Day 1 to Day 10 (total duration: max. 10 days).
Part B - Multiple ascending dose (MAD): t½ after last dose administration. | Blood samples for the determination of the PK parameters will be collected at predefined time points from Day 1 to Day 10 (total duration: max. 10 days).

CONTACTS AND LOCATIONS:
Locations (1):
- Parexel International GmbH Klinikum Westend, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No